CLINICAL TRIAL: NCT00173433
Title: The Importance of Exogenous Reinfection in the Tuberculosis Endemic of Taiwan
Brief Title: Exogenous Reinfection of Tuberculosis in Taiwan
Status: Completed | Type: Observational
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 9461700627
Record Dates: First submitted 2005-09-12; First posted 2005-09-15 (Estimated); Last update posted 2014-12-09 (Estimated); Status verified 2014-12

CONDITIONS: Tuberculosis
Keywords: tuberculosis; relapse; reinfection; reactivation; dormancy; tuberculin skin test
MeSH Terms: conditions — Tuberculosis; Recurrence; Reinfection

GROUPS / COHORTS (1):
- Culture-confirmed relapse of TB: Patients who have a recurrent episode of culture-confirmed TB after completion of treatment for the first episode of culture-confirmed TB

SUMMARY:
we hypothesize that exogenous reinfection is very important in the Taiwan endemic. Therefore, we design a series of studies to evaluate the individual contribution of exogenous reinfection and endogenous reactivation in the Taiwan endemic, and to realize the impact of exogenous reinfection. First, we will identify the patients with TB relapse after complete treatment. The M. tuberculosis isolates responsible for their initial and recurrent episodes will then be genotyped to clarify the percentage of exogenous reinfection and endogenous reinfection.

DETAILED DESCRIPTION:
Tuberculosis (TB) remains the most important infectious disease in the world. In Taiwan, the incidence of TB increased in recent years. The failure of control implies the necessity to reevaluate the epidemiology of Mycobacterium tuberculosis. It is widely thought that most cases of TB are caused by reactivation of a latent infection. Treatment programs have therefore focused on cure rates rather than tracking of additional cases. But recent studies showed that exogenous reinfection plays an important role in the development of TB. In addition, it seems that the higher the local incidence, the more important exogenous reinfection is. The question of exogenous reinfection versus endogenous reactivation has an impact on the distribution of resources for the prevention and treatment of TB. Based on these evidences, we hypothesize that exogenous reinfection is very important in the Taiwan endemic. Therefore, we design a series of studies to evaluate the individual contribution of exogenous reinfection and endogenous reactivation in the Taiwan endemic, and to realize the impact of exogenous reinfection. First, we will identify the patients with TB relapse after complete treatment. The M. tuberculosis isolates responsible for their initial and recurrent episodes will then be genotyped to clarify the percentage of exogenous reinfection and endogenous reinfection.

ELIGIBILITY:
Inclusion Criteria:

* culture-proven tuberculosis with recurrence

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2005-08; Primary Completion 2006-07 (Actual); Study Completion 2006-07 (Actual)

PRIMARY OUTCOMES:
relapse due to reinfection | 6 years
  proportion of patients with exogenous reinfection in those with relapse of TB

CONTACTS AND LOCATIONS:
Overall Officials: Jann-Yuan Wang, MD, Principal Investigator — National Taiwan University Hospital
Locations (1):
- National Taiwan University Hospital, Taipei, Taiwan

REFERENCES:
- [Background] Bandera A, Gori A, Catozzi L, Degli Esposti A, Marchetti G, Molteni C, Ferrario G, Codecasa L, Penati V, Matteelli A, Franzetti F. Molecular epidemiology study of exogenous reinfection in an area with a low incidence of tuberculosis. J Clin Microbiol. 2001 Jun;39(6):2213-8. doi: 10.1128/JCM.39.6.2213-2218.2001. PMID 11376059
- [Background] Behr MA, Warren SA, Salamon H, Hopewell PC, Ponce de Leon A, Daley CL, Small PM. Transmission of Mycobacterium tuberculosis from patients smear-negative for acid-fast bacilli. Lancet. 1999 Feb 6;353(9151):444-9. doi: 10.1016/s0140-6736(98)03406-0. PMID 9989714
- [Background] Blumberg HM, Burman WJ, Chaisson RE, Daley CL, Etkind SC, Friedman LN, Fujiwara P, Grzemska M, Hopewell PC, Iseman MD, Jasmer RM, Koppaka V, Menzies RI, O'Brien RJ, Reves RR, Reichman LB, Simone PM, Starke JR, Vernon AA; American Thoracic Society, Centers for Disease Control and Prevention and the Infectious Diseases Society. American Thoracic Society/Centers for Disease Control and Prevention/Infectious Diseases Society of America: treatment of tuberculosis. Am J Respir Crit Care Med. 2003 Feb 15;167(4):603-62. doi: 10.1164/rccm.167.4.603. No abstract available. PMID 12588714
- [Background] Caminero JA, Pena MJ, Campos-Herrero MI, Rodriguez JC, Afonso O, Martin C, Pavon JM, Torres MJ, Burgos M, Cabrera P, Small PM, Enarson DA. Exogenous reinfection with tuberculosis on a European island with a moderate incidence of disease. Am J Respir Crit Care Med. 2001 Mar;163(3 Pt 1):717-20. doi: 10.1164/ajrccm.163.3.2003070. PMID 11254530
- [Background] Caminero JA, Pena MJ, Campos-Herrero MI, Rodriguez JC, Garcia I, Cabrera P, Lafoz C, Samper S, Takiff H, Afonso O, Pavon JM, Torres MJ, van Soolingen D, Enarson DA, Martin C. Epidemiological evidence of the spread of a Mycobacterium tuberculosis strain of the Beijing genotype on Gran Canaria Island. Am J Respir Crit Care Med. 2001 Oct 1;164(7):1165-70. doi: 10.1164/ajrccm.164.7.2101031. PMID 11673204
- [Background] Cronin WA, Golub JE, Lathan MJ, Mukasa LN, Hooper N, Razeq JH, Baruch NG, Mulcahy D, Benjamin WH, Magder LS, Strickland GT, Bishai WR. Molecular epidemiology of tuberculosis in a low- to moderate-incidence state: are contact investigations enough? Emerg Infect Dis. 2002 Nov;8(11):1271-9. doi: 10.3201/eid0811.020261. PMID 12453355
- [Background] Davies BH. Infectivity of tuberculosis. Thorax. 1980 Jul;35(7):481-2. doi: 10.1136/thx.35.7.481. No abstract available. PMID 7434308
- [Background] Ellis BA, Crawford JT, Braden CR, McNabb SJ, Moore M, Kammerer S; National Tuberculosis Genotyping and Surveillance Network Work Group. Molecular epidemiology of tuberculosis in a sentinel surveillance population. Emerg Infect Dis. 2002 Nov;8(11):1197-209. doi: 10.3201/eid0811.020403. PMID 12453343
- [Background] Garbe TR, Hibler NS, Deretic V. Isoniazid induces expression of the antigen 85 complex in Mycobacterium tuberculosis. Antimicrob Agents Chemother. 1996 Jul;40(7):1754-6. doi: 10.1128/AAC.40.7.1754. PMID 8807080
- [Background] Garcia de Viedma D, Marin M, Hernangomez S, Diaz M, Ruiz Serrano MJ, Alcala L, Bouza E. Tuberculosis recurrences: reinfection plays a role in a population whose clinical/epidemiological characteristics do not favor reinfection. Arch Intern Med. 2002 Sep 9;162(16):1873-9. doi: 10.1001/archinte.162.16.1873. PMID 12196086
- [Background] Glassroth J, Robins AG, Snider DE Jr. Tuberculosis in the 1980s. N Engl J Med. 1980 Jun 26;302(26):1441-50. doi: 10.1056/NEJM198006263022603. No abstract available. PMID 6990260
- [Background] Jou NT, Yoshimori RB, Mason GR, Louie JS, Liebling MR. Single-tube, nested, reverse transcriptase PCR for detection of viable Mycobacterium tuberculosis. J Clin Microbiol. 1997 May;35(5):1161-5. doi: 10.1128/jcm.35.5.1161-1165.1997. PMID 9114400
- [Background] Miller AC, Sharnprapai S, Suruki R, Corkren E, Nardell EA, Driscoll JR, McGarry M, Taber H, Etkind S. Impact of genotyping of Mycobacterium tuberculosis on public health practice in Massachusetts. Emerg Infect Dis. 2002 Nov;8(11):1285-9. doi: 10.3201/eid0811.020316. PMID 12453357
- [Background] Pai SR, Actor JK, Sepulveda E, Hunter RL Jr, Jagannath C. Identification of viable and non-viable Mycobacterium tuberculosis in mouse organs by directed RT-PCR for antigen 85B mRNA. Microb Pathog. 2000 Jun;28(6):335-42. doi: 10.1006/mpat.2000.0353. PMID 10839970
- [Background] Sharnprapai S, Miller AC, Suruki R, Corkren E, Etkind S, Driscoll J, McGarry M, Nardell E. Genotyping analyses of tuberculosis cases in U.S.- and foreign-born Massachusetts residents. Emerg Infect Dis. 2002 Nov;8(11):1239-45. doi: 10.3201/eid0811.020370. PMID 12453348
- [Background] Sokolove PE, Mackey D, Wiles J, Lewis RJ. Exposure of emergency department personnel to tuberculosis: PPD testing during an epidemic in the community. Ann Emerg Med. 1994 Sep;24(3):418-21. doi: 10.1016/s0196-0644(94)70178-4. PMID 8080139
- [Background] Stead WW. Management of health care workers after inadvertent exposure to tuberculosis: a guide for the use of preventive therapy. Ann Intern Med. 1995 Jun 15;122(12):906-12. doi: 10.7326/0003-4819-122-12-199506150-00003. PMID 7755225
- [Background] Supply P, Mazars E, Lesjean S, Vincent V, Gicquel B, Locht C. Variable human minisatellite-like regions in the Mycobacterium tuberculosis genome. Mol Microbiol. 2000 May;36(3):762-71. doi: 10.1046/j.1365-2958.2000.01905.x. PMID 10844663
- [Background] van Embden JD, Cave MD, Crawford JT, Dale JW, Eisenach KD, Gicquel B, Hermans P, Martin C, McAdam R, Shinnick TM, et al. Strain identification of Mycobacterium tuberculosis by DNA fingerprinting: recommendations for a standardized methodology. J Clin Microbiol. 1993 Feb;31(2):406-9. doi: 10.1128/jcm.31.2.406-409.1993. PMID 8381814
- [Background] van Rie A, Warren R, Richardson M, Victor TC, Gie RP, Enarson DA, Beyers N, van Helden PD. Exogenous reinfection as a cause of recurrent tuberculosis after curative treatment. N Engl J Med. 1999 Oct 14;341(16):1174-9. doi: 10.1056/NEJM199910143411602. PMID 10519895